CLINICAL TRIAL: NCT02565277
Title: The Effect of Influenza Vaccination on the Systemic Inflammatory Response and Myocardial Protection in Patients Undergoing Cardiac Surgery: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Health Sciences North Research Institute (Other)
Responsible Party: Principal Investigator, Rony Atoui, Msc, MD, FRCSC, Cardiac Surgeon, Health Sciences North Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AMRIC Dr.Atoui
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Systemic Inflammatory Response
MeSH Terms: interventions — Influenza Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza Vaccine (Active Comparator): Fluzone injection once IM
  Interventions: Biological: Influenza Vaccine
- Placebo (Placebo Comparator): Saline Injection once IM
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Influenza Vaccine
  Other Names: Fluzone
  Arms: Influenza Vaccine
Drug: Placebo
  Other Names: Saline Injection
  Arms: Placebo

SUMMARY:
To assess the impact of influenza vaccination on the overall systemic inflammatory response in patients undergoing cardiac surgery and investigate functional and clinical outcomes in vaccinated patients postoperatively.

DETAILED DESCRIPTION:
The investigators propose to perform a single center, double-blind, randomized, placebo-controlled crossover trial analyzing the beneficial effect of the influenza vaccine in patients undergoing cardiac surgery. This study assesses the impact of the influenza vaccination on the overall systemic inflammatory response and investigates the functional and clinical outcome in vaccinated patients after cardiac surgery. The study sample will consist of patients undergoing cardiac surgery at Health Sciences North randomized into 2 groups: 1) those who receive the vaccine or placebo preoperatively, or: 2) those who receive the vaccine or placebo 4-6 weeks postoperatively. Subjects in both groups will be compared using standard laboratory tools to assess the level of various pro- and anti-inflammatory cytokines (IL-6, IL-8,TNF-alpha, IL-10) as well as other cardiac and inflammatory markers (troponins, CRP), at different time intervals intra- and post-operatively. Other clinical outcomes will also be collected prospectively and compared between the 2 groups. These include hemodynamic parameters as well as major postoperative events. Further assessments will include the Frailty Index and Scale (in patients 65+) and length of stay after surgery

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol (i.e. return for follow-up visits, and able to converse with study personnel)
* Age 18 years or older
* Undergoing major cardiac surgery using cardiopulmonary bypass

Exclusion Criteria:

* Have not received influenza vaccination in the past or cannot be vaccinated due to previous severe reaction to influenza vaccine, egg, latex, or thimerosol allergies, or refusal of vaccination
* Participant has received a community available influenza vaccine within <6 months
* History of Guillain-Barré syndrome
* Immunosuppressive disorders or medications (including oral prednisone >10 mg daily, recent chemotherapy treatment)
* Emergency cases as determined by the investigator or physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Pro and anti-inflammatory cytokines and inflammatory markers | Nine Months

CONTACTS AND LOCATIONS:
Overall Officials: Roni Atoui, MSc MD FRCSC, Principal Investigator — Health Sciences North Research Institute
Locations (1):
- Health Sciences North Research Institute, Greater Sudbury, Ontario, Canada